CLINICAL TRIAL: NCT00817791
Title: Phase 1 Study of Protective Effect of Hyperbaric Oxygen Preconditioning on Brain and Myocardium Injury During CABG Surgery
Brief Title: Preconditioning With Hyperbaric Oxygen in Cardiovascular Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: LZXiong,YLi, Department of Anaesthesiology,Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: liyang2007
Record Dates: First submitted 2009-01-02; First posted 2009-01-06 (Estimated); Last update posted 2009-06-15 (Estimated); Status verified 2009-03

CONDITIONS: Brain Injury; Myocardial Injury
Keywords: CABG; hyperbaric oxygen; preconditioning; S100B; NSE; Troponin I; CABG surgery; neuroprotection
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HBO (Experimental)
  Interventions: Device: Hyperbaric oxygen pretreatment (GR2200)

INTERVENTIONS:
Device: Hyperbaric oxygen pretreatment (GR2200) — 2 hours/day,5 days before surgery
  Other Names: GR2200

SUMMARY:
Animal studies have shown that preconditioning with hyperbaric oxygen can induce central nervous system and heart ischemic tolerance. This study was designed to determine the protective effect of hyperbaric oxygen preconditioning on brain and myocardium ischemia-reperfusion injury during coronary artery bypass graft surgery.

DETAILED DESCRIPTION:
60 patients scheduled to undergo coronary revascularization were recruited for this trial. Exclusion criteria included Emergency operation, age older than 80 years, learning difficulty, previous cerebrovascular disease, visual or hearing impairment, history of pneumothorax, Claustrophobia, middle ear disease, EF < 35%. Patients were randomized either to the control group or hyperbaric oxygen group. The laboratory analysis of markers included S100B, NSE and troponin I. The assessment of cognitive dysfunction was performed 5 days before surgery and 7 days after surgery and haemodynamic measurements, length of stay in ICU, length of stay in hospital post-operation were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo coronary revascularization surgery.

Exclusion Criteria:

* Emergency operation
* Age older than 80 years
* Learning difficulty
* Previous cerebrovascular disease
* Visual or hearing impairment
* History of pneumothorax, claustrophobia, middle ear disease, EF < 35%

Max Age: 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2007-11; Primary Completion 2008-08 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Post operative cognitive dysfunction | 5 days before surgery and 7 days after surgery

SECONDARY OUTCOMES:
S100B protein,NSE and Troponin I | Within the first 3 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: xiong L Z, doctor, Study Chair — Department of anaesthiology,Xijing hospital